CLINICAL TRIAL: NCT00949975
Title: A 12-week, Randomised, Double-blind, Placebo-controlled, Parallel Group, Multinational, Phase IIb Dose Range Finding Study to Evaluate the Efficacy and Safety of AZD9668 Administered Orally at 3 Dose Levels to Patients With Chronic Obstructive Pulmonary Disease (COPD) on Treatment With Tiotropium
Brief Title: A Dose Range Finding Study to Evaluate the Efficacy and Safety of AZD9668 Administered Orally at Three Dose Levels to Patients With Chronic Obstructive Pulmonary Disease (COPD) on Treatment With Tiotropium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0520C00012
Record Dates: First submitted 2009-07-21; First posted 2009-07-31 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic; Obstructive; Pulmonary; Lung; Respiratory disease; Efficacy; Safety and tolerability; Placebo-controlled; Pharmacokinetics; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Respiration Disorders | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): AZD9668 active treatment
  Interventions: Drug: AZD9668
- 2 (Active Comparator): AZD9668 active treatment
  Interventions: Drug: AZD9668
- 3 (Active Comparator): AZD9668 active treatment
  Interventions: Drug: AZD9668
- 4 (Placebo Comparator): AZD9668 placebo treatment
  Interventions: Drug: AZD9668 Placebo

INTERVENTIONS:
Drug: AZD9668 — 2 x 30 mg oral tablets twice daily (bid) for 12 weeks
  Arms: 1
Drug: AZD9668 — 2 x 10 mg oral tablets twice daily (bid) for 12 weeks
  Arms: 2
Drug: AZD9668 — 2 x 2.5 mg oral tablets twice daily (bid) for 12 weeks
  Arms: 3
Drug: AZD9668 Placebo — 2 x Matched placebo to oral tablet twice daily (bid) for 12 weeks
  Arms: 4

SUMMARY:
The primary objective is to evaluate the dose-response relationship and efficacy of AZD9668 at 3 dose levels compared with placebo in symptomatic COPD patients by assessing effects on lung function and symptoms of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with symptoms over 1 year
* Smokers or ex-smokers
* Males or post-menopausal females between 40 and 80 years old
* Able to use electronic devices

Exclusion Criteria:

* Past history or current evidence of clinically significant heart disease
* Current diagnosis of asthma
* Patients who require long term oxygen therapy
* Treatment with antibiotics within 4 weeks of study visit 1b

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Volgemeier, Dr., Principal Investigator — Director der Klinik fur Innere Medizin mit Schwerpunkt Pneumologie-Universitatsklinikum GieBen und Marburg, D-35043 Marburg, Germany
Locations (105):
- United States (9):
  - Research Site, Fullerton, California
  - Research Site, Valparaiso, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Hickory, North Carolina
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
- Australia (8):
  - Research Site, Concord, New South Wales
  - Research Site, Glebe, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Daw Park, South Australia
  - Research Site, Parkville, Victoria
  - Research Site, Nedlands, Western Australia
- Canada (14):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, Antigonish, Nova Scotia
  - Research Site, Grimsby, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, La Malbaie, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Germany (5):
  - Research Site, Berlin
  - Research Site, Fulda
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Marburg
- Japan (24):
  - Research Site, Seto, Aichi-ken
  - Research Site, Noda, Chiba
  - Research Site, Touon, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Yukuhashi, Fukuoka
  - Research Site, Nihommatsu, Fukushima
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Himeji, Hyōgo
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Ukyo-ku, Kyoto, Kyoto
  - Research Site, Matsumoto, Nagano
  - Research Site, Saiki, Oita Prefecture
  - Research Site, Kishiwada, Osaka
  - Research Site, Kita-ku, Sakai, Osaka
  - Research Site, Matsue, Shimane
  - Research Site, Chūō, Tokyo
  - Research Site, Nakano-ku, Tokyo
  - Research Site, Tanabe, Wakayama
  - Research Site, Bunkyō City
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa City, Batangas
  - Research Site, Quezon City
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Chęciny
  - Research Site, Krakow
  - Research Site, Ostrów Wielkopolski
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Tczew
  - Research Site, Wroclaw
  - Research Site, Zawadzkie
- Russia (6):
  - Research Site, Barnaul, Russia
  - Research Site, Kazan', Russia
  - Research Site, Moscow, Russia
  - Research Site, Novosibirsk, Russia
  - Research Site, Saint Petersburg, Russia
  - Research Site, Yekaterinburg, Russia
- Slovakia (11):
  - Research Site, Bardejov
  - Research Site, Bojnice
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Trnava
  - Research Site, Zvolen
  - Research Site, Žilina
- South Korea (6):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Uijeongbu-si, Gyeonggi-do
  - Research Site, Anyang
  - Research Site, Bucheon-si
  - Research Site, Daegu
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Ukraine (5):
  - Research Site, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Research Site, Luhansk, Ukraine
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv

REFERENCES:
- [Derived] Leidy NK, Murray LT, Monz BU, Nelsen L, Goldman M, Jones PW, Dansie EJ, Sethi S. Measuring respiratory symptoms of COPD: performance of the EXACT- Respiratory Symptoms Tool (E-RS) in three clinical trials. Respir Res. 2014 Oct 7;15(1):124. doi: 10.1186/s12931-014-0124-z. PMID 25287629
- [Derived] Leidy NK, Murray LT, Jones P, Sethi S. Performance of the EXAcerbations of chronic pulmonary disease tool patient-reported outcome measure in three clinical trials of chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Mar;11(3):316-25. doi: 10.1513/AnnalsATS.201309-305OC. PMID 24432712
- [Derived] Vogelmeier C, Aquino TO, O'Brien CD, Perrett J, Gunawardena KA. A randomised, placebo-controlled, dose-finding study of AZD9668, an oral inhibitor of neutrophil elastase, in patients with chronic obstructive pulmonary disease treated with tiotropium. COPD. 2012 Apr;9(2):111-20. doi: 10.3109/15412555.2011.641803. PMID 22458939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 13 July 2009. Last patient completed 05 August 2010. Study conducted at 138 centres in 12 countries (Australia, Canada, Germany, Japan, Korea, Philippines, Poland, Russia, Slovakia, Taiwan, Ukraine and US)
Pre-assignment Details: Patients were stabilised on maintenance therapy (tiotropium, 18 micrograms od) during a 2-week run-in period before randomisation.
Groups:
- 5 mg AZD9668: AZD9668 2x2.5 mg oral tablets twice daily (bid) for 12 weeks
- 20 mg AZD9668: AZD9668 2x10 mg oral tablets twice daily (bid) for 12 weeks
- 60 mg AZD9668: AZD9668 2x30 mg oral tablets twice daily (bid) for 12 weeks
- Placebo: Matched Placebo Tablets
Period: Overall Study
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Started | 212 | 206 | 202 | 218
Completed | 185 | 177 | 183 | 190
Not Completed | 27 | 29 | 19 | 28
Not completed — Voluntary discontinuation | 6 | 5 | 3 | 6
Not completed — Adverse Event | 11 | 11 | 10 | 10
Not completed — Safety reason | 0 | 1 | 0 | 0
Not completed — Study-specific criteria | 0 | 1 | 1 | 0
Not completed — Incorrect enrolment | 5 | 10 | 4 | 7
Not completed — Severe non-compliance | 3 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 3
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo | Total
Number analyzed (Participants) | 212 | 206 | 202 | 218 | 838
Age Continuous [Mean (Full Range); unit: Years] | 62 [42 to 80] | 63 [42 to 79] | 61 [40 to 79] | 62 [41 to 80] | 62 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 53 | 53 | 199
  Male | 166 | 159 | 149 | 165 | 639

OUTCOME MEASURES:

1. Primary Outcome: Baseline Pre-bronchodilator FEV1 (L)
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: The efficacy analysis set for each outcome measure includes those patients who received at least one dose of investigational product and for whom a baseline and at least one post-randomisation measurement is available for that outcome measure. Patients were analysed by to randomised treatment in accordance with the intention to treat principle.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 201 | 216
L | 1.51 (0.471) | 1.47 (0.468) | 1.50 (0.512) | 1.51 (0.467)

2. Primary Outcome: End-value Pre-bronchodilator FEV1 (L)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 201 | 216
L | 1.51 (0.018) [lower limit 0.018] | 1.47 (0.018) [lower limit 0.018] | 1.46 (0.018) [lower limit 0.018] | 1.47 (0.018) [lower limit 0.018]

3. Secondary Outcome: Post-bronchodilator FEV1 (L) - Baseline
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 199 | 201 | 215
L | 1.68 (0.501) | 1.64 (0.472) | 1.65 (0.516) | 1.69 (0.471)

4. Secondary Outcome: Post-bronchodilator FEV1 (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 199 | 201 | 215
L | 1.66 (0.017) [lower limit 0.017] | 1.63 (0.017) [lower limit 0.017] | 1.63 (0.017) [lower limit 0.017] | 1.62 (0.017) [lower limit 0.017]

5. Secondary Outcome: Pre-bronchodilator FVC (L) - Baseline
Description: Forced Vital Capacity (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 201 | 216
L | 3.08 (0.850) | 3.01 (0.739) | 3.06 (0.856) | 3.04 (0.754)

6. Secondary Outcome: Pre-bronchodilator FVC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 201 | 216
L | 3.08 (0.026) [lower limit 0.026] | 3.05 (0.026) [lower limit 0.026] | 3.02 (0.026) [lower limit 0.026] | 3.02 (0.025) [lower limit 0.025]

7. Secondary Outcome: Post-bronchodilator FVC (L) - Baseline
Description: Forced Vital Capacity (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 199 | 201 | 215
L | 3.30 (0.914) | 3.24 (0.723) | 3.24 (0.885) | 3.27 (0.781)

8. Secondary Outcome: Post-bronchodilator FVC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 199 | 201 | 215
L | 3.28 (0.023) [lower limit 0.023] | 3.26 (0.024) [lower limit 0.024] | 3.24 (0.024) [lower limit 0.024] | 3.22 (0.023) [lower limit 0.023]

9. Secondary Outcome: Pre-bronchodilator IC (L) - Baseline
Description: Inspiratory Capacity (L) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 200 | 216
L | 2.22 (0.680) | 2.14 (0.563) | 2.15 (0.662) | 2.17 (0.574)

10. Secondary Outcome: Pre-bronchodilator IC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 199 | 200 | 216
L | 2.15 (0.027) [lower limit 0.027] | 2.15 (0.028) [lower limit 0.028] | 2.16 (0.027) [lower limit 0.027] | 2.15 (0.026) [lower limit 0.026]

11. Secondary Outcome: Post-bronchodilator IC (L) - Baseline
Description: Inspiratory Capacity (L) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 206 | 199 | 201 | 214
L | 2.37 (0.709) | 2.30 (0.601) | 2.28 (0.677) | 2.32 (0.628)

12. Secondary Outcome: Post-bronchodilator IC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: Measured at clinic visits: 1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 206 | 199 | 201 | 214
L | 2.29 (0.025) [lower limit 0.025] | 2.30 (0.025) [lower limit 0.025] | 2.31 (0.025) [lower limit 0.025] | 2.30 (0.025) [lower limit 0.025]

13. Secondary Outcome: PEF - Baseline Measured by Patient at Home (L/Min) in the Morning
Description: Peak Expiratory Flow (L/min) as a measure of lung function, measured at home by the patient each morning.Baseline is the mean of last 10 days of data before start of treatment
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
L/min | 222.33 (83.177) | 219.86 (90.395) | 216.99 (91.299) | 221.79 (89.005)

14. Secondary Outcome: PEF - End-value Measured by Patient at Home (L/Min) in the Morning
Description: Peak Expiratory Flow (L/min)
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
L/min | 214.30 (2.899) [lower limit 2.899] | 214.55 (2.920) [lower limit 2.920] | 212.35 (2.944) [lower limit 2.944] | 220.47 (2.840) [lower limit 2.840]

15. Secondary Outcome: FEV1 - Baseline Measured by Patient at Home (L) in the Morning
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured at home by the patient each morning.Baseline is the mean of last 10 days of data before start of treatment
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
L | 1.40 (0.521) | 1.34 (0.444) | 1.36 (0.507) | 1.38 (0.456)

16. Secondary Outcome: FEV1 - End-value Measured by Patient at Home (L) in the Morning
Description: Forced Expiratory Volume in 1 second (L)
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
L | 1.36 (0.018) [lower limit 0.018] | 1.35 (0.018) [lower limit 0.018] | 1.33 (0.018) [lower limit 0.018] | 1.34 (0.018) [lower limit 0.018]

17. Secondary Outcome: EXACT - Baseline Total Score
Description: EXAcerbations of Chronic pulmonary disease Tool, patient questionnaire as a measure of respiratory symptoms (reported as units on a 0 (best health status) to 100 (worst possible status)scale). Baseline is the mean of last 10 days of data before start of treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 205 | 200 | 214
Units on a scale | 43.17 (10.109) | 42.38 (8.166) | 42.37 (9.320) | 40.95 (9.725)

18. Secondary Outcome: EXACT - End-value Total Score
Description: EXAcerbations of Chronic pulmonary disease Tool, patient questionnaire as a measure of respiratory symptoms (reported as units on a 0 (best health status) to 100 (worst possible status)scale). Last 6 weeks on treatment.
Time Frame: Measured daily in the evening for 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 207 | 205 | 200 | 214
Units on a scale | 39.97 (0.545) [lower limit 0.545] | 39.72 (0.543) [lower limit 0.543] | 40.59 (0.552) [lower limit 0.552] | 39.71 (0.533) [lower limit 0.533]

19. Secondary Outcome: BCSS - Baseline Total Score
Description: Breathlessness, Cough and Sputum Scale, patient reported questionnaire as a measure of respiratory symptoms (reported on a 0 (best health status) to 12 (worst possible status)scale).Baseline is the mean of last 10 days of data before start of treatment
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
Units on a scale | 4.85 (1.954) | 4.66 (1.526) | 4.79 (1.756) | 4.48 (1.782)

20. Secondary Outcome: BCSS - End-value Total Score
Description: Breathlessness, Cough and Sputum Scale, patient reported questionnaire as a measure of respiratory symptoms (reported on a 0(best health status) to 12(worst possible status)scale). Last 6 weeks on treatment
Time Frame: Measured daily in the evening for 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 217
Units on a scale | 4.09 (0.098) [lower limit 0.098] | 4.03 (0.099) [lower limit 0.099] | 4.25 (0.100) [lower limit 0.100] | 4.20 (0.096) [lower limit 0.096]

21. Secondary Outcome: Sputum Colour - Baseline
Description: Sputum Colour as assessed by the Bronkotest scale, reported on a scale from 1 - clear (best health status) to 5 - dark green (worst possible health status).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 194 | 179 | 188 | 195
Units on a scale | 2.15 (1.069) | 2.34 (1.137) | 2.13 (0.956) | 2.16 (1.046)

22. Secondary Outcome: Sputum Colour - End Value
Description: Sputum Colour as assessed by the Bronkotest scale, reported on a scale from 1 - clear (best health status) to 5 - dark green (worst possible health status).End of treatment week 12
Time Frame: Measured at clinic visits:1, 4, 8 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 194 | 179 | 188 | 195
Units on a scale | 2.11 (0.062) [lower limit 0.062] | 2.03 (0.065) [lower limit 0.065] | 2.20 (0.063) [lower limit 0.063] | 2.11 (0.062) [lower limit 0.062]

23. Secondary Outcome: Use of Reliever Medication
Description: Daily average of number of inhalations of reliever medication
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Inhalations
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 209 | 204 | 202 | 215
Inhalations | 4.28 (0.173) [lower limit 0.173] | 4.20 (0.175) [lower limit 0.175] | 4.65 (0.175) [lower limit 0.175] | 4.56 (0.170) [lower limit 0.170]

24. Secondary Outcome: Six-minute Walk Test - Distance Walked at Baseline (m)
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 194 | 184 | 191 | 205
m | 386.2 (125.22) | 402.2 (111.98) | 384.9 (115.50) | 386.0 (132.48)

25. Secondary Outcome: Six-minute Walk Test - End-value Distance Walked (m)
Description: distance walked on vist 6 - last on treatment clinic visit
Time Frame: Measured Day 1 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: m
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 194 | 184 | 191 | 205
m | 396.7 (4.74) [lower limit 4.74] | 397.8 (4.87) [lower limit 4.87] | 411.2 (4.76) [lower limit 4.76] | 409.5 (4.61) [lower limit 4.61]

26. Secondary Outcome: St George's Respiratory Questionnaire (COPD) - Overall Score at Baseline
Description: St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease, as a measure of Quality of Life (reported on a % scale from 0 (best health status) to 100(worst possible status)).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 199 | 187 | 194 | 210
Scores on a scale | 53.98 (18.276) | 51.98 (18.207) | 52.97 (18.234) | 51.41 (18.849)

27. Secondary Outcome: St George's Respiratory Questionnaire (COPD) - End-value Overall Score
Description: St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease, as a measure of Quality of Life (reported on a % scale from 0 (best health status) to 100(worst possible status)).questionaire assessed on vist 6 -( last on treatment clinic visit)
Time Frame: Measured Day 1 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 199 | 187 | 194 | 210
Scores on a scale | 49.50 (1.014) [lower limit 1.014] | 49.49 (1.049) [lower limit 1.049] | 47.93 (1.023) [lower limit 1.023] | 46.35 (0.984) [lower limit 0.984]

28. Secondary Outcome: Exacerbations - Clinic Defined
Description: Number of patients having a clinic defined disease exacerbation
Time Frame: Duration of the the treatment period - 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 210 | 205 | 202 | 218
Participants | 29 | 28 | 34 | 29

ADVERSE EVENTS:
Arm/Group | 5 mg AZD9668 | 20 mg AZD9668 | 60 mg AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 7/212 | 14/206 | 15/202 | 9/218
Other Adverse Events (participants affected / at risk) | 17/212 | 14/206 | 13/202 | 24/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg AZD9668 (N=212) | 20 mg AZD9668 (N=206) | 60 mg AZD9668 (N=202) | Placebo (N=218)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROINTESTINAL ULCER HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 2 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 7 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
'RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg AZD9668 (N=212) | 20 mg AZD9668 (N=206) | 60 mg AZD9668 (N=202) | Placebo (N=218)
NASOPHARYNGITIS (Infections and infestations) | 15 | 9 | 9 | 13
HEADACHE (Nervous system disorders) | 3 | 5 | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No